CLINICAL TRIAL: NCT07160426
Title: Pilot Study of Protection And Repair of Endothelial-glycocalyx in Sepsis (SPARES)
Brief Title: Study of Protection And Repair of Endothelial-glycocalyx in Sepsis
Acronym: SPARES
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: University of Colorado Health (Other)
Responsible Party: Principal Investigator, Nathan Shapiro, Professor of Emergency Medicine, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPARES Pilot
Record Dates: First submitted 2025-08-29; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Sepsis
Keywords: Sepsis; Fresh Frozen Plasma; Endothelium; glycocalyx
MeSH Terms: conditions — Sepsis | interventions — Ringer's Lactate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Experimental: FFP Bolus (Experimental): Two-unit initial FFP bolus, then one unit every 12 hours for 48 hours (total 5 units).
  Interventions: Biological: Fresh Frozen Plasma (blood product)
- Experimental: FFP Continuous Infusion (Experimental): 5 units FFP infused continuously at ~42 mL/hr over 48 hours.
  Interventions: Biological: Fresh Frozen Plasma (blood product)
- Placebo Comparator: Lactated Ringer's + Multivitamins (Placebo Comparator): Placebo given as either (a) 500 mL LR bolus, then 250 mL q12h for 48h (total 1,250 mL), or (b) 500 mL over 12h, repeated to total 2,000 mL over 48h; prepared by pharmacy to match plasma appearance.
  Interventions: Drug: MVI and lactated ringers

INTERVENTIONS:
Biological: Fresh Frozen Plasma (blood product) — Fresh Frozen Plasma
  Arms: Experimental: FFP Bolus; Experimental: FFP Continuous Infusion
Drug: MVI and lactated ringers — placebo
  Arms: Placebo Comparator: Lactated Ringer's + Multivitamins

SUMMARY:
Sepsis damages the blood vessel lining and its protective "glycocalyx," contributing to organ failure and death. This pilot, randomized, blinded study will test whether giving fresh frozen plasma (FFP)-either as intermittent boluses or as a continuous infusion-protects or repairs the glycocalyx compared with look-alike placebo fluid (lactated Ringer's with multivitamins), and whether this leads to better clinical outcomes. We will measure blood and urine biomarkers of glycocalyx injury and track organ support needs, ICU/hospital-free days, and survival through 28-90 days.

DETAILED DESCRIPTION:
Multicenter, blinded, placebo-controlled randomized pilot trial comparing: (1) FFP bolus regimen; (2) FFP continuous infusion; and (3) placebo (LR with multivitamins, administered as bolus or continuous to maintain blinding). Primary biologic readout is change in syndecan-1 (glycocalyx degradation) with additional endothelial activation and inflammation markers; key clinical endpoints include mortality and organ failure-free days. Target enrollment is 45 adults with sepsis (SOFA ≥2) within ICU or ED settings.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Confirmed or suspected infection (pathogen detected or antimicrobial administered)
* SOFA score ≥2
* ICU patient or ED patient with anticipated ICU admission

Exclusion Criteria:

* Unable to randomize within 24h of meeting inclusion criteria
* Current hospitalization >2 days
* Decision to withhold life-sustaining treatment (exception for DNR only)
* Moribund; not expected to survive 24h
* Life expectancy <28 days from non-sepsis condition
* Any condition where participation isn't in the patient's best interest or limits assessments
* Prisoner
* Pregnancy
* Concurrent interventional trial with overlapping treatments/outcomes
* Inability to obtain patient/LAR consent
* History of Transfusion Related Acute Lung Injury (TRALI) or Transfusion Associated Circulatory Overload (TACO)
* End Stage Renal Disease
* Chronic tracheostomy with ventilator use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Syndecan-1 | baseline to study days 1,3,5
  Syndecan-1 measurement

SECONDARY OUTCOMES:
All-cause mortality to Day 28 | 28 days
  All-cause mortality to Day 28
Organ failure-free days | 28 days
  Organ failure-free days to Day 28 (alive and without assisted ventilation, new RRT, or vasopressors).
SOFA Score | change over days 1, 3, 5
  SOFA score

IPD SHARING:
Plan to Share IPD: Undecided
Will depend on scientific merit